CLINICAL TRIAL: NCT00305786
Title: Phase II Study of Oxaliplatin in Combination With Gemcitabine for 2 Line Treatment of NSCLC Patients With Advanced and Metastatic Disease
Brief Title: Gemcitabine and Oxaliplatin as Second-Line Therapy in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20043597; SCCC-2004078 (Other: University of Miami Institutional Review Board); WIRB-20050485 (Other: Western Institutional Review Board)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with oxaliplatin works as second-line therapy in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy and safety of gemcitabine hydrochloride and oxaliplatin as second-line chemotherapy in patients with stage IIIB or IV non-small cell lung cancer.
* Determine overall response in patients treated with this regimen.

Secondary

* Determine time to progression, time to treatment failure, and overall survival of these patients.
* Determine the type, frequency, severity, timing, and relatedness of all adverse events during treatment and for 30 days after completion of study treatment.
* Assess the quality of life of these patients.
* Determine the expression of RRM1 and ERCC1 in peripheral blood mononuclear cells from these patients.

OUTLINE: This is an open-label, nonrandomized study.

Patients receive gemcitabine hydrochloride IV over 100 minutes followed by oxaliplatin IV over 2 hours on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at the beginning of each course, at the completion of study treatment, and then every 6 weeks thereafter.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IIIB or IV non-small cell lung cancer (NSCLC)
* Failed first-line chemotherapy

  * Must have received ≥ 1, but no more than 2, prior chemotherapy regimens for stage IIIB or IV NSCLC

    * Prior radiotherapy or surgery for earlier stage disease allowed, provided target lesions chosen for response assessment have not have been irradiated
* At least 1 unidimensionally measurable lesion with diameter ≥ 20 mm by conventional methods OR ≥ 10 mm by spiral CT scan

  * If a single lesion is identified as the target lesion, histological or cytological confirmation of this lesion is required
* No symptomatic brain metastases

  * Clinically stable brain metastases on a stable dose of (or no longer requiring) dexamethasone allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver involvement)
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after completion of study treatment
* No history of an acute cardiac or CNS event within the past 6 months, including any of the following:

  * Unstable angina
  * Myocardial infarction
  * Clinically relevant arrhythmia
  * Stroke
* No current clinical evidence of congestive heart failure or unstable coronary artery disease
* No peripheral neuropathy > grade 1
* No history of hypersensitivity to study drugs
* No serious uncontrolled medical or psychiatric illness, including any of the following:

  * Serious infection
  * Interstitial pneumonia
  * Extensive and symptomatic fibrosis of the lung
* No other malignancy within the past year, except for squamous cell or basal cell carcinoma of the skin, carcinoma in situ of the cervix, or superficial transitional cell carcinoma of the bladder

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior surgery
* At least 4 weeks since prior cranial radiation for brain metastases
* More than 4 weeks since prior participation in another investigational drug study
* No concurrent immunotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by RECIST criteria | At study completion

SECONDARY OUTCOMES:
Toxicity as monitored by DSMC | At study completion

CONTACTS AND LOCATIONS:
Overall Officials: Caio Max S. Rocha Lima, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida